CLINICAL TRIAL: NCT04922268
Title: External Focus of Attention Feedback to Mitigate Posttraumatic Osteoarthritis Risk After ACL Reconstruction
Brief Title: External Focus of Attention Posttraumatic Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Abbey Thomas, PhD, Assistant Professor, University of North Carolina, Charlotte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-0089
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear; Osteo Arthritis Knee
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internal focus of attention feedback (Active Comparator): Participants will complete 12 sessions over 3 weeks receiving visual feedback in a mirror of their movement patterns.
  Interventions: Other: Internal focus of attention feedback
- External focus of attention feedback (Experimental): Participants will complete 12 sessions over 3 weeks receiving visual feedback of their movement patterns from a laser.
  Interventions: Other: External focus of attention feedback

INTERVENTIONS:
Other: Internal focus of attention feedback — Participants will complete 12 sessions over a 3-week period of functional movement retraining while receiving mirror feedback. Participants will be instructed to perform each functional task in a manner that keeps their knee in line with their toes.
  Arms: Internal focus of attention feedback
Other: External focus of attention feedback — Participants will complete 12 sessions over a 3-week period of functional movement retraining while receiving visual feedback via laser. Participants will be instructed to perform each functional task in a manner that does causes the laser to move up and down but not side-to-side.
  Arms: External focus of attention feedback

SUMMARY:
Knee injuries, especially those to the ACL, are common among physically active people. These injuries are frequently treated with surgical reconstruction (ACL reconstruction; ACLR). While ACLR restores stability it does not protect against future injury, long-term pain, disability, and arthritis associated with these injuries. Our study is going to examine new ways to provide feedback about the way people move to determine if these are better at modifying movement patterns that are known risk factors of posttraumatic osteoarthritis development than current standard treatments. If you participate, you will be asked to undergo a movement analysis in a research laboratory while you perform tasks such as walking and hopping. After this initial assessment, you will be randomly allocated to one of 2 treatment groups. Each treatment group will perform 4 weeks (3x/week) of exercises to change the way people walk. Participants will then report for follow-up movement analysis testing 1- and 4-weeks after completing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* history of primary, unilateral ACL reconstruction 6-24 months prior to enrollment
* cleared to return to full activity by treating orthopedic surgeon

Exclusion Criteria:

* Body mass index >35 kg/m2
* History of musculoskeletal injury sustained 3 months prior to enrollment
* Current participation in formal post-operative rehabilitation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in lower extremity biomechanics during walking | 1-week post-intervention, 4-weeks post-intervention
  Knee and hip angles and loads measured via 3D biomechanics
Knee cartilage health | 1-week post-intervention, 4-weeks post-intervention
  Knee cartilage thickness measured using diagnostic ultrasound imaging

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No